CLINICAL TRIAL: NCT01760603
Title: A Prospective,Multicenter Pilot Study to Evaluate the Clinical Performance of the Ischia Spinous Fascia Fixation Surgery for Pelvic Organ Prolapse.
Brief Title: Ischia Spinous Fascia Fixation Surgery for Pelvic Organ Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pumch-gyn-04
Record Dates: First submitted 2012-12-25; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ISFF (Experimental): The patients performed ischia spinous fascia fixation surgery.
  Interventions: Procedure: ISFF

INTERVENTIONS:
Procedure: ISFF — Ischia spinous fascia fixation surgery was performed on patient with pelvic organ prolapse.

SUMMARY:
Pelvic organ prolapse is a common problem. The primary treatment is surgery. Ischia spinous fascia fixation procedure is developed in China for vaginal apex fixation with native tissue.

This study is designed to determine the effectiveness and safety of ischia spinous fascia fixation procedure for the treatment of pelvic organ prolapse stage III.

Patients enrolled into the study will be followed up for up to 3 years after surgery. Evaluation will take place during surgery and postoperative visit. Stage of prolapse before and after surgery, patient satisfaction through quality of life and sexual function questionnaires before and after surgery, and peri-operative complication rates will be evaluated.

DETAILED DESCRIPTION:
Pelvic Organ prolapse (a feeling of bulge in the vagina) may cause some distressing symptoms such as loss of control of the bowel or bladder, and may also cause problems with patient's sex life. An ideal procedure for vaginal apical support should provide a durable suspension, have minimal complications, and not affect sexual or visceral function.

Ischia spinous fascia fixation procedure is developed in China. It is a transvaginal procedure used for restoring the vaginal apex support with native tissue. Clinical practice showed that it was safe, efficient and cost-effective. Recurrent rate after 1 year follow-up was about 10%, and quality of life improved significantly from the baseline.

The purpose of this multicenter, prospective study is to evaluate the effectiveness and safety of this procedure in the treatment of symptomatic pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Candidates with symptomatic pelvic organ prolapse of POP-Q Stage II or more, suitable for surgical repair.
* Vaginal hysterectomy and anti-incontinence procedures could be performed concurrently.
* Agrees to participate in the study, including completion of all study-related procedures, evaluations and questionnaires.

Exclusion Criteria:

* Previous repair of pelvic organ prolapse involving insertion of mesh.
* Experimental drug or experimental medical device within 3 months prior to the planned procedure.
* Active genital, urinary or systemic infection at the time of the surgical procedure. Surgery may be delayed in such subjects until the infection is cleared.
* Coagulation disorder or on therapeutic anticoagulant therapy at the time of surgery.
* History of chemotherapy or pelvic radiation therapy.
* Systemic disease known to affect bladder or bowel function (e.g. Parkinson's disease, multiple sclerosis, spinal cord injury or trauma).
* Current evaluation or treatment for chronic pelvic pain (e.g. interstitial cystitis, endometriosis, coccydynia, vulvodynia).
* Nursing or pregnant or intends future pregnancy.
* Chronic cough not well-controlled.
* BMI ≥ 30.
* In the investigator's opinion, any medical condition or psychiatric illness that could potentially be life threatening or affect their ability to complete the study visits according to this protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Anatomical improvement according to POP-Q Score | 6 weeks
Anatomical improvement according to POP-Q Score | 1 year
Anatomical improvement according to POP-Q Score | 2 years
Anatomical improvement according to POP-Q Score | 3 years

SECONDARY OUTCOMES:
Hospital data including operative time, estimated blood loss, length of stay, postoperative mortality, time of voiding recovery | At discharge, an expected average of 5 days after operation

OTHER OUTCOMES:
Presence/absence of complications (composite score) | Up to 6 weeks
  The occurrence (in the per-operative phase or within 6 weeks post-op) of at least one of the following: 1) bleeding complications; 2) infectious complications; 3) any wound caused by a surgeon movement: bladder, ureteral, or vascular injuries; 4)medical complications: deep vein thrombosis, pulmonary embolism and etc.Complications will be categorized using the Dindo surgical complication grading scale
Change from baseline in PFIQ-7 scores | 6 month, 1 year, 2 years and 3 years
n subjects sexually active at baseline, assessment of sexual function using PISQ-12 (mean scores and change from baseline) | 6 months, 1 year, 2 years and 3 years
Subject global impression assessed on a 5 point Likert scale | 6 months, 1 year, 2 years, 3 years
Presence/absence of complications (composite score) | up to 3 years
  Long-term negative outcomes of the surgical procedure will also be recorded until 3 years after surgery. For example, de novo urinary incontinence, de novo dyspareunia and overall failure rate. Complications will be categorized using the Dindo surgical complication grading scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, Principal Investigator — Peking Union Medical College Hospital
Locations (4):
- China (4):
  - Foshan Maternal and Child Health Hospital, Foshan, Guangdong
  - The third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Affiliated Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Peking Union Medical College Hospital, Beijing